CLINICAL TRIAL: NCT05900505
Title: Addressing Child and Family Social Determinants of Health Needs With Social Navigation: Navigating Social Resources for Children's Health "NSRCH" Clinic
Brief Title: Social Navigator to Address Social Determinants of Health in Pediatrics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Caroline Zuijdwijk, Pediatric Endocrinologist, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22/65X
Record Dates: First submitted 2023-04-19; First posted 2023-06-12 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will be referred to a social navigator to address their identified social needs.
  Interventions: Other: Social Navigator
- Control Group (No Intervention): Participants in the control group will be referred to a social worker, as per standard care.

INTERVENTIONS:
Other: Social Navigator — The social navigator will assess patient/family needs and help them to access community resources (specific to their community) to address these, while promoting their engagement and self-efficacy.
  Arms: Intervention Group

SUMMARY:
It is crucial to understand the social and economic context in which children and youth live; their social determinants of health (SDH). Although this is well recognized, many health care providers do not address SDH because of the lack of easily accessible resources once social needs are identified.

Social workers (SW) have the ability to support families once a social need has been identified. However, not every clinic has a SW, and even those that do often struggle to meet the needs of all the families requiring support.

The use of social navigators (SN) is an innovative solution for an unmet need. SN models have been successful in primary care settings, but, to date, have not been adapted to address the SDH needs of children and their families receiving care in pediatric specialty care settings. We will implement the first of its kind pediatric SN clinic at the Children's Hospital of Eastern Ontario (CHEO): "Navigating Social Resources for Children's Health" (NSRCH). Our study will evaluate NSRCH - an innovative, transferable, and low-cost pediatric-specific SN model. Our goal is to support families with SDH needs to access timely, appropriate supports and resources via NSRCH.

DETAILED DESCRIPTION:
In Phase 1 of our study, potential patient-participants will be identified from the type 1 diabetes and type 2 diabetes clinics at CHEO in the following way: the study coordinator will manually screen upcoming patients in the diabetes clinic schedules in Epic. Then, a cover letter and study information sheet will be sent to potential patient-participants (or they would be approached by a study coordinator in-person during the clinic visit). They will follow up with the family to explain the study, answer any questions, confirm interest. Interested families will be asked to complete the Phase 1 Screening Tool.

The study coordinator will be automatically notified of all positive screens (at least 1 identified social need), and then contact the respective families to invite them to participate in Phase 2 of the study and obtain informed consent.

At baseline, the coordinator will collect baseline data and have the families complete the Quality of Life - Brief Version (WHOQOL-BREF) and Baseline Questionnaire. After the visit, participants will be randomized to the intervention or control groups using the randomization module in REDCap. A referral will then be forwarded to either the SN or SW. All clinic visits between baseline and follow up will be scheduled directly by the SN or SW. The SN and the SW will be asked to complete a checklist for each participant consultation, and the results will be summarized by the coordinator.

Participants will be contacted by a coordinator for a follow up visit at 6 months. At which time, they will collect follow-up data and have the families complete the Phase 1 Screening Tool, WHOQOL-BREF, and CSQ.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

* Parent or guardian of a child, aged between 0-17 years
* Parent or guardian of a patient in the T1D or T2D clinics at CHEO

Phase 2

* Parent or guardian of a child, aged between 0-17 years
* Parent or guardian of a patient in the T1D or T2D clinics at CHEO
* At least 1 positive response on the SDH Phase 1 Screening Tool
* Optional: child consented to allow access to medical information via electronic medical chart

Exclusion Criteria:

* Active social work client at the time of administration of the Phase 1 Screening Tool, defined as families who have had active follow up with a diabetes SW within the last 3 months, with plans for ongoing follow up.
* Unable or unwilling to provide i) implied consent for the completion of the SDH Phase 1 Screening Tool and/or ii) written informed consent for participation in the Phase 2 randomized trial

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To compare participant satisfaction with NSRCH (social navigator) vs. standard care (social worker), as measured by the Client Satisfaction Questionnaire (CSQ). | 6 months
  Client Satisfaction Questionnaire: Participant satisfaction will be determined using a validated Client Satisfaction Questionnaire (CSQ). The CSQ is scored on a scale of 8 to 32, with higher scores indicating higher satisfaction.

SECONDARY OUTCOMES:
To compare the time to access NSRCH (social navigator) vs. standard care (social worker). | 6 months
To compare the rate of attendance to NSRCH (social navigator) vs. standard care (social worker) visits. | 6 months
To compare the number of community resources accessed by participants relative to the number of community resources to which they were referred by NSRCH (social navigator) vs. standard care (social worker). | 6 months
To compare whether resources provided to the participants corresponded to their identified social needs at NSRCH (social navigator) vs. standard care (social worker). | 6 months
  The social workers and social navigator will be required to indicate which resources were referred to each participant. They will also be required to indicate if the resource corresponds to one or more of the participant's identified social need(s). The mean percentage of resources that correspond to identified social needs will be compared between NSRCH (social navigator) and standard care (social workers).
To compare change in Quality of Life (QOL) of participants (pre/post intervention) referred to NSRCH (social navigator) vs standard care (social worker), as measured by the WHOQOL-BREF. | 6 months
  Quality of Life: change in quality of life from baseline to end of study (pre/post intervention) will be compared between the NSRCH and standard care groups. Quality of life will be assessed using the World Health Organization Quality of Life - Brief Version (WHOQOL-BREF). The WHOQOL-BREF is a quality of life assessment developed by the WHOQOL Group with fifteen international field centres, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally. Higher scores denote a higher quality of life. This measure provides 4 domain scores, one for each domain in which quality of life is assessed: physical (raw score 7-35), psychological (raw score 6-30), social relationships (raw score 3-15), and environment (raw score 8-40). Raw scores can also be transformed to reflect scores of 4-20 or 0-100.

OTHER OUTCOMES:
To compare NSRCH (social navigator) vs. standard care (social worker) with respect to changes in glycemic control. | 6 months
  To compare NSRCH (social navigator) vs. standard care (social worker) with respect to changes in glycemic control: Glycated hemoglobin (HbA1c, (%)), percent time in range (TIR - percentage of time in previous 14 days spent within target glucose range of 70-180 mg/dL or 3.9-10 mmol/L), and glucose management indicator (GMI, %). Taken together, these indicators reflect overall glycemic control.
Change in Social Determinants of Health (SDH) Screening Status | 6 months
  To compare the change in positive screen status on the SDH screening tool from baseline to 6 months, in NSRCH (social navigator) vs. standard care (social worker).
To compare the resource cost of the social navigator compared to the social worker. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Zuijdwijk, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario - Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT05900505/ICF_000.pdf